CLINICAL TRIAL: NCT04726410
Title: Cold Stored Platelet Early Intervention in Traumatic Brain Injury Trial
Brief Title: Cold-stored Platelet Early Intervention in TBI
Acronym: CriSP-TBI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jason Sperry (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Jason Sperry, Professor of Surgery and Critical Care Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY20070044; W81XWH-16-D-0024 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2021-01-12; First posted 2021-01-27 (Actual); Results first posted 2025-04-29 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Cold Stored Platelets
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: permuted block design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cold-stored Platelet (CSP) (Experimental): early infusion of up to 2 units of urgent release cold stored platelets (CSP)
  Interventions: Biological: Cold Stored Platelets
- Standard care (Active Comparator): standard care therapy
  Interventions: Biological: Standard Care

INTERVENTIONS:
Biological: Cold Stored Platelets — early infusion of urgent release CSP
  Arms: Cold-stored Platelet (CSP)
Biological: Standard Care — standard care including room temperature platelets
  Arms: Standard care

SUMMARY:
The Cold Stored Platelet Early Intervention in Traumatic Brain Injury (CriSP-TBI) trial is a proposed 3 year, open label, single center, randomized trial designed to determine the feasibility, efficacy, and safety of urgent release cold stored platelets (CSP) in patients with TBI requiring platelet transfusion. Patients will be randomized to receive either standard care or early infusion of urgent release cold stored platelets (CSP). The proposed pilot study will enroll at the University of Pittsburgh and will enroll approximately 100 patients. The primary outcome for the pilot trial is feasibility, with principal secondary clinical outcome of 6-month Extended Glasgow Outcome Scale (GOS-E).

DETAILED DESCRIPTION:
Platelet transfusion is commonly provided to patients with moderate or severe TBI who are on antiplatelet medications. Evidence suggests that patients on antiplatelet medications may have worse outcomes following TBI. Current literature has not demonstrated major outcome improvements in those patients who receive platelet transfusion. This lack of significant benefit may be due to insufficient dosing or due to the poor hemostatic function of standard care room temperature platelets. Studying the potential benefits of Cold Stored Platelet transfusion in the TBI population will provide needed direct comparison of room temperature and cold stored platelet transfusion which is unable to occur in patients with hemorrhagic shock, who may require large volumes of red blood cells and plasma concomitantly with platelet transfusion.

By providing Cold Stored Platelets in an urgent release fashion following injury, a potentially superior hemostatic agent is given early, closer to the time of injury. The current pilot trial was designed to determine the feasibility, efficacy and safety of urgent release cold stored platelets as compared to standard care in TBI patients requiring platelet transfusion. There are no high-level data which appropriately characterize the urgent release use of cold stored platelets out to 14 days or their function over that time period as compared to standard room temperature platelets. These results will be able to inform future large randomized clinical trials allowing the most appropriate injured population, inclusion criteria, and primary outcome to be selected and utilized.

ELIGIBILITY:
Inclusion Criteria:

Patients with traumatic brain injury, defined by presence of potential progressive intracranial injury on CT scan, at significant risk for urgent neurosurgical procedure as determined by neurosurgical evaluation, who meet at least one of the following:

1. History or indication of pre-injury antiplatelet agent use
2. Need for platelet transfusion per standard practice

Exclusion Criteria:

1. Wearing NO CriSP opt out bracelet
2. Hypotension in Emergency Department (SBP< 90 mmHg)
3. Age > 89 or < 18 years of age
4. Penetrating injury
5. Prisoner
6. Pregnancy
7. Going to operating room for non-neurosurgical intervention in first 60 minutes
8. Platelet transfusion contraindications per care team (for example, recent vascular stent, embolic stroke, intracranial and/or vascular lesions)
9. Objection to study voiced by participant or family member in Emergency Department
10. Currently on therapeutic anticoagulant in addition to aspirin and/or clopidogrel (e.g. warfarin, direct-acting oral anticoagulants)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason L Sperry, MD, Study Director — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with the funding agency as well as other researchers upon request to the Investigational New Drug (IND) Sponsor and Principal Investigator.
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available after publication of the primary manuscript
Access Criteria: Requests for data will be submitted in writing and reviewed by the IND Sponsor and Principal Investigator

REFERENCES:
- [Derived] Brunskill SJ, Disegna A, Wong H, Fabes J, Desborough MJ, Doree C, Davenport R, Curry N, Stanworth SJ. Blood transfusion strategies for major bleeding in trauma. Cochrane Database Syst Rev. 2025 Apr 24;4(4):CD012635. doi: 10.1002/14651858.CD012635.pub2. PMID 40271704

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cold-stored Platelet (CSP) | Standard Care
Started | 50 | 50
Completed | 50 | 49
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cold-stored Platelet (CSP) | Standard Care | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 73.5 [67 to 80] | 78 [66 to 82] | 76 [66 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 47
  Male | 27 | 26 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 44 | 37 | 81
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 7 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Study Feasibility
Description: proportion of eligible patients that can be randomized, enrolled, adhere to protocol, and complete follow-up
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cold-stored Platelet (CSP) | Standard Care
Number analyzed (Participants) | 50 | 50
Participants | 50 | 50

2. Secondary Outcome: 6-month Extended Glasgow Outcome Scale (GOS-E)
Description: A tool used to characterize 6-month functional status into 8 defined categories, with 1 being the worst (death) to 8 being the most favorable (good recovery).
Time Frame: 6 months after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Cold-stored Platelet (CSP) | Standard Care
Number analyzed (Participants) | 43 | 40
Participants
  Unfavorable | 21 | 20
  Favorable | 22 | 20

3. Secondary Outcome: 24-hour Mortality
Description: Mortality within 24 hours
Time Frame: Enrollment through 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Cold-stored Platelet (CSP) | Standard Care
Number analyzed (Participants) | 50 | 49
Participants | 1 | 0

4. Secondary Outcome: In-hospital Mortality
Description: Mortality in-hospital
Time Frame: Enrollment through discharge up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cold-stored Platelet (CSP) | Standard Care
Number analyzed (Participants) | 50 | 49
Participants | 6 | 7

5. Secondary Outcome: TBI Progression
Description: Evidence of progression of TBI. Common Data Elements for CT scan indicators of TBI progression will be utilized.
Time Frame: Enrollment through 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Cold-stored Platelet (CSP) | Standard Care
Number analyzed (Participants) | 48 | 47
Participants | 8 | 11

6. Secondary Outcome: Galveston Orientation and Amnesia Test (GOAT)
Description: 10-item questionnaire used to quickly assess post-traumatic amnesia following head injury. The GOAT is read orally to the patient and may be easily administered at the bedside. The total score accounts for orientation of person, place, and time, and recollection of events pre and post- injury. Cutoff scores are available to identify abnormal, borderline, and normal orientation. The total GOAT score is obtained by deducting the sum of the error points from each incorrect response from 100.Range is 0-100. A score of 66 or lower is categorized as "impaired," 66-75 as "borderline," and 76-100 as "normal." This will be obtained At Discharge from Current Hospital Admission
Time Frame: At Discharge from Current Hospital Admission
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cold-stored Platelet (CSP) | Standard Care
Number analyzed (Participants) | 38 | 36
score on a scale | 95 [72 to 100] | 91 [71 to 100]

7. Secondary Outcome: Incidence of Allergic/Transfusion Reaction
Description: Any transfusion complication in Emergency Department or Operating Room
Time Frame: Enrollment through 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Cold-stored Platelet (CSP) | Standard Care
Number analyzed (Participants) | 50 | 49
Participants | 0 | 0

8. Secondary Outcome: Incidence of Transfusion Related Acute Lung Injury (TRALI)
Description: Occurrence of Acute Respiratory Distress Syndrome (ARDS) within 6 hours of transfusion of platelets
Time Frame: Enrollment through 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Cold-stored Platelet (CSP) | Standard Care
Number analyzed (Participants) | 50 | 49
Participants | 0 | 0

9. Secondary Outcome: Incidence of Thromboembolic Events
Description: Incidence of pulmonary embolism, venous thrombosis, or arterial thrombosis
Time Frame: Enrollment through 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Cold-stored Platelet (CSP) | Standard Care
Number analyzed (Participants) | 50 | 49
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Cold-stored Platelet (CSP) | Standard Care
All-Cause Mortality (participants affected / at risk) | 6/50 | 7/49
Serious Adverse Events (participants affected / at risk) | 9/50 | 8/49
Other Adverse Events (participants affected / at risk) | 0/50 | 0/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cold-stored Platelet (CSP) (N=50) | Standard Care (N=49)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
pulmonary consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
seizures (Nervous system disorders) | 0 (0) | 1 (1)
deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1)
other (Infections and infestations) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-08): https://cdn.clinicaltrials.gov/large-docs/10/NCT04726410/Prot_SAP_001.pdf
  • Informed Consent Form (2023-10-03): https://cdn.clinicaltrials.gov/large-docs/10/NCT04726410/ICF_000.pdf